CLINICAL TRIAL: NCT02427594
Title: Acid-Base Compensation in Chronic Kidney Disease: Measurement and Physiologic Impact
Brief Title: Acid-Base Compensation in Chronic Kidney Disease
Acronym: ABC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Pro00058905; K23DK095949 (NIH)
Record Dates: First submitted 2015-04-23; First posted 2015-04-28 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-04

CONDITIONS: Chronic Kidney Disease
Keywords: Kidney Diseases; Renal Insufficiency, Chronic; Dietary nonvolatile acid load; Blood pressure; Urine net acid excretion
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Diseases | interventions — Sodium Bicarbonate; baking powder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Controlled diet first (Experimental): In this arm participants will first consume a controlled diet plus added table salt (sodium chloride) for one week. They will then consume an identical controlled diet plus sodium bicarbonate for one week. Sodium bicarbonate will be dosed as 2,600 mg divided three times daily if ideal body weight is <70 kg or 3,250 mg divided three times daily if ideal body weight is ≥70 kg. Added table salt will match the sodium content of the sodium bicarbonate dose (i.e. 31 or 39 mEq/day).
  Interventions: Drug: Sodium bicarbonate; Other: Controlled diet
- Sodium bicarbonate first (Experimental): In this arm participants will first consume a controlled diet plus sodium bicarbonate for one week. They will then consume an identical controlled diet plus added table salt (sodium chloride) for one week. Sodium bicarbonate will be dosed as 2,600 mg divided three times daily if ideal body weight is <70 kg or 3,250 mg divided three times daily if ideal body weight is ≥70 kg. Added table salt will match the sodium content of the sodium bicarbonate dose (i.e. 31 or 39 mEq/day).
  Interventions: Drug: Sodium bicarbonate; Other: Controlled diet

INTERVENTIONS:
Drug: Sodium bicarbonate — Drug/dietary supplement is used in a crossover design to lower the nonvolatile acid load of the diet compared to the control period.
  Other Names: Baking powder
Other: Controlled diet — Diet without sodium bicarbonate supplementation

SUMMARY:
The purpose of this study is to evaluate changes in urine net acid excretion, blood pressure and body chemistry that occur when the dietary acid load is lowered by using a drug/dietary supplement similar to baking soda. This may be important for patients with kidney disease because they may have difficulty removing all of the dietary acid load from the body in the urine. Participants with and without kidney disease will be recruited. Each participant will be fed a controlled diet for one week with sodium bicarbonate and for one week without sodium bicarbonate to evaluate these changes. The investigators will also determine if the effect of dietary acid load reduction is different in patients with kidney disease compared to those without kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* estimated glomerular filtration rate ≥30 ml/min/1.73m2
* serum bicarbonate 20-28 mEq/L

Exclusion Criteria:

* diabetes mellitus
* uncontrolled hypertension or recent (<3 weeks) titration of blood pressure medications
* clinically significant volume overload on screening physical examination
* selected medical conditions other than kidney disease and hypertension (active cancer, chronic liver failure, moderate to severe COPD, New York Heart Association class 2 or greater congestive heart failure, obstructive sleep apnea requiring nightly continuous positive airway pressure, solid organ transplant)
* use of alkali supplementation
* body mass index <18.5 or >40 kg/m2
* ideal body weight <45.5 kg
* anemia at screening (hematocrit <29% in participants with kidney disease or <33% in healthy participants)
* pregnancy or breastfeeding
* allergies, intolerance or unwillingness to consume foods or supplement provided in feeding menu
* serum calcium less than 8.6 mg/dl on screening laboratories

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-04; Primary Completion 2017-08-25 (Actual); Study Completion 2017-08-25 (Actual)

PRIMARY OUTCOMES:
Change in ambulatory blood pressure | Measured at the end of each week of intervention (i.e. one week apart)
  Change in mean 24 hour systolic and diastolic blood pressure comparing the end of the controlled feeding plus sodium bicarbonate period to the end of the controlled feeding plus table salt period.
Change in urine net acid excretion | Urine net acid excretion will be measured at three timepoints over approximately 3 weeks (i.e. 2 weeks of intervention plus one week baseline data collection/run-in)
  Change in urine net acid excretion comparing the end of the controlled feeding plus sodium bicarbonate period to the end of the controlled feeding plus table salt period.

SECONDARY OUTCOMES:
Change in clinic blood pressure | Clinic blood pressure will be measured at multiple timepoints over approximately 3 weeks (i.e. 2 weeks of intervention plus one week baseline data collection/run-in)
  Change in average of three readings of systolic and diastolic blood pressure will be evaluated comparing the end of the controlled feeding plus sodium bicarbonate period to the end of the controlled feeding plus table salt period.
Change in plasma nitric oxide metabolites | Measured at the end of each week of intervention (i.e. one week apart) up to 3 weeks
  Change in nitric oxide metabolites comparing the end of the controlled feeding plus sodium bicarbonate period to the end of the controlled feeding plus table salt period.

OTHER OUTCOMES:
Differences in metabolomic profiles | Measured at the end of each week of intervention (i.e. one week apart) up to 3 weeks
  Differences in metabolites will be evaluated comparing the end of the controlled feeding plus sodium bicarbonate period to the end of the controlled feeding plus table salt period.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Scialla, Principal Investigator — Duke University
Locations (1):
- Duke University School of Medicine, Durham, North Carolina, United States

REFERENCES:
- [Derived] Tyson CC, Luciano A, Modliszewski JL, Corcoran DL, Bain JR, Muehlbauer M, Ilkayeva O, Pourafshar S, Allen J, Bowman C, Gung J, Asplin JR, Pendergast J, Svetkey LP, Lin PH, Scialla JJ. Effect of Bicarbonate on Net Acid Excretion, Blood Pressure, and Metabolism in Patients With and Without CKD: The Acid Base Compensation in CKD Study. Am J Kidney Dis. 2021 Jul;78(1):38-47. doi: 10.1053/j.ajkd.2020.10.015. Epub 2021 Mar 31. PMID 33810868